CLINICAL TRIAL: NCT07305961
Title: Studio Nazionale Sull'Epidemiologia ed Efficacia Delle Terapie Nel Trattamento Della Scabbia
Brief Title: National Study on the Epidemiology and Effectiveness of Therapies in the Treatment of Scabies
Acronym: SCAB-net
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Other Study IDs: SID06; RSO ID - 477 (Other: AIFA)
Record Dates: First submitted 2025-06-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective cohort: Patients diagnosed with scabies who attend outpatient clinics and their close contacts (household members and partners) at the various participating centres from the date of study approval until 31/12/2025 will be included, along with additional parameters regarding treatment, failures and epidemiological and clinical assessments.
  Interventions: Other: data collection
- retrospective cohort: Only the number of registered scabies cases and the presence or absence of treatment failures will be considered; no clinical patient data will be extrapolated.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Biographical data: age; immunodeficiency; bedridden condition. Household data: number of people in the household, original state of the household, presence of paediatric cases weighing more or less than 15 kg, presence of a language barrier.
  Diagnostic criteria: clinical, dermatoscopic and/or microscopic. Clinical data: affected areas, non-specific therapies previously carried out. Days of isolation of the index case (if applicable). Treatment data: the first specific anti-mite therapy carried out, including the mode of administration; the number of days since the onset of the illness; the number of people treated per index case; the drug with which recovery was achieved (if known); and the time taken for recovery. Data for investigating treatment failures: answers to questions concerning treatment carried out with close contacts and cohabitants, correct information about environmental remediation implementation, number of therapy cycles carried out and follow-up timeframe.
  Groups: prospective cohort
Other: data collection — Only the number of registered scabies cases and whether or not treatment has failed will be taken into account. No clinical data from the patients will be extrapolated.
  Groups: retrospective cohort

SUMMARY:
Multicentre retrospective, prospective, non-profit, national observational study

DETAILED DESCRIPTION:
Scabies is an infectious skin condition caused by the mite Sarcoptes scabiei var. hominis. This mite can only parasitise and reproduce in the outermost layer of human skin (the stratum corneum). The disease is typically transmitted through human-to-human contact, though it can also be transmitted through fomites. It affects between 200 and 300 million people worldwide each year, with considerable variation in prevalence ranging from 0.2% to 71.4% in different regions. Over the past 10-20 years, the frequency of epidemics appears to be increasing, not only in countries where scabies is prevalent, but also in states that have historically experienced low rates of infection.The increase in cases across Europe, coupled with the rapid epidemic spread of the disease and the emergence of resistance to topical treatments, underscores the imperative for a comprehensive and systematic study involving multiple centres.

The primary guidelines for managing scabies involve performing environmental hygiene measures, such as washing and changing clothing daily and cleaning all surfaces that come into contact with the skin.

In terms of treatment, the European Society of Dermatology and Venereology guidelines recommend topical permethrin or benzyl benzoate and oral ivermectin as first-line treatments.

Apply topical permethrin 5% cream in the evening to cool, dry skin all over your body, including the folds, navel, limbs, genitals, the area behind your ears and under your nails. If there are any suspicious lesions, the scalp and face should also be treated, avoiding the areas around the eyes and lips. Leave the cream in place for 8-12 hours and apply a second dose after 7-14 days.

Oral ivermectin should be taken as a single dose at a dosage of 200 μg/kg, repeated in the same manner after seven days. Although European guidelines recommend taking it on a full stomach, the manufacturer and other guidelines recommend taking it on an empty stomach.

Benzyl benzoate lotion at a concentration of 10-25% is applied for two evenings and left in place for 8-12 hours. A third application should be made after seven days.

The treatment should be carried out not only by the patient, but also by their close contacts - usually members of their household - and should be extended to anyone who has had prolonged and continuous contact with individuals who are ill.

Topical permethrin cream at 5% is the first-line treatment for scabies in Italy. However, there has recently been an increase in reports of treatment failure. This phenomenon has also become increasingly prevalent in many other European countries. Therapy failure is likely to be due to a combination of factors, including drug resistance. Incorrect use of the treatment in terms of the amount of active ingredient, the method of application and/or the timing could be the cause of treatment failure.

The increase in cases in Europe, the rapid spread of the disease and the growing phenomenon of treatment resistance highlight the need for a large, systematic study involving several centres. Therefore, we propose a national multicentre retrospective and prospective observational study that aims to evaluate epidemiological data (prevalence, incidence, affected ethnicities and population groups), the most frequently used treatments, and treatment failures.

This study aims to evaluate the success rate of first-line therapies according to European guidelines in patients diagnosed with scabies and their close contacts (family members/caregivers). This will be achieved by observing patients with scabies who attend outpatient clinics for diagnosis, treatment and/or follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with clinical and/or dermoscopic and/or microscopic diagnosis of scabies.
* Close contacts (household/relatives) of patients diagnosed with scabies.
* Obtaining informed consent.

Exclusion Criteria:

* There are no exclusion criteria.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with scabies and their close contacts (household/partners) afferent to the outpatient clinics of participating Italian centers during the duration of the study will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1332 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | From the date of enrolment until the date of healing, assessed up to 52 weeks.
  The cure rate is represented by the number of patients who were cured after the first treatment.

SECONDARY OUTCOMES:
Frequency of scabies diagnosis | From the date of enrolment to the previous three years
  Assess the trend in the absolute frequency of scabies diagnoses over the past three years.
Epidemiological analyses | at the end of the study
  Conduct descriptive epidemiological analyses by categorising the observed cases according to age group, ethnicity, and time distribution over the study period.
body distribution | Baseline
  Evaluate which body areas are most affected by the disease, and establish whether involvement in certain areas predicts treatment failure.
presence/absence of clinical parameters | Baseline
  Evaluate the clinical parameters of the index case, such as immunodepression and allurement. Consider whether any previous non-specific therapies may have increased the likelihood of treatment failure.
presence/absence of language barriers | Baseline
  Evaluate whether a language barrier exists between healthcare workers and patients, as incorrect intake of therapy in terms of dosage and timing, as well as a lack of or incorrect environmental hygiene measures, may be correlated with treatment failure or re-infestation.

CONTACTS AND LOCATIONS:
Locations (1):
- APSS - Ospedale Santa Chiara, Trento, Italy/Trento, Italy